CLINICAL TRIAL: NCT04425590
Title: The Role of DLBS1033 in the Management of Acute Ischemic Stroke Patients: Study Protocol for a Randomized Controlled Study
Brief Title: The Benefit of Add On DLBS1033 for Ischemic Stroke Patient
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Duta Wacana Christian University (Other)
Collaborators: Dexa Laboratories Of Biomolecular Science (Unknown)
Responsible Party: Principal Investigator, Rizaldy Taslim Pinzon, Principal investigator, Neurologist, Duta Wacana Christian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INADLBS
Record Dates: First submitted 2020-05-27; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Ischemic Stroke
Keywords: DLBS1033; Standard therapy; Stroke; Outcomes; Lumbrokinase
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — DLBS 1033; Aspirin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Vitamin B 12

STUDY DESIGN:
Intervention Model Description: Eligible subjects were randomly allocated to receive any of the following regiments: standard therapy consists of aspirin 100 mg once daily, atorvastatin 20 mg once daily, vitamin B12 100 mg three times daily (control group) or standard therapy and DLBS1033 3 times daily (experimental group).
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): standard therapy consists of aspirin 100 mg once daily, atorvastatin 20 mg once daily, vitamin B12 100 mg three times daily and DLBS1033 3 times daily (experimental group).
  Interventions: Drug: DLBS1033; Drug: Aspirin; Drug: Statin; Drug: Vit B12
- Control Group (Active Comparator): standard therapy consists of aspirin 100 mg once daily, atorvastatin 20 mg once daily, vitamin B12 100 mg three times daily
  Interventions: Drug: Aspirin; Drug: Statin; Drug: Vit B12

INTERVENTIONS:
Drug: DLBS1033 — DLBS 1033 490 mg tablet 3 times daily
  Other Names: Disolf
  Arms: Experimental Group
Drug: Aspirin — Aspirin 100 mg tablet once daily
Drug: Statin — Atorvastatin 20 mg tablet once daily
  Other Names: Atorvastatin
Drug: Vit B12 — Vit B12 100 mg tablet three times daily

SUMMARY:
Stroke is one of the most common non-communicable diseases worldwide. It is the leading cause of morbidity and mortality in many countries.

Stroke is broadly classified into ischemic and hemorrhagic stroke. Ischemic stroke is more common than hemorrhagic stroke. In Indonesia, the prevalence of ischemic stroke is 42.9% compare to hemorrhagic stroke 19.9%. Ischemic stroke defined as an episode of neurological dysfunction caused by focal cerebral, spinal, or retinal infarction.

One of the main therapy in ischemic stroke is administration of anti thrombotic agent. DLBS1033 is a bioactive protein fraction isolated from Lumbricus rubellus. DLBS1033 possessed quadruple activities that inhibit platelet aggregation, induces fibrinogenolysis, fibrinolysis, and thrombolysis. This is a new proposed medication nowadays. There is still a limited study about DLBS1033. To our knowledge, research concern on the usage of DLBS1033 in stroke patients is very limited in Indonesia. This study aimed to Measure the benefit of DLBS1033 as add on therapy for ischemic stroke patients.

The hypothesis of this study :

a. The use of DLBS1033 improve functional status of ischemic stroke patients at hospital discharge. b. The use of DLBS1033 improve functional status 30-days after stroke onset.

DETAILED DESCRIPTION:
This was randomized, controlled, open-label, study from the period of April 2020 - August 2020 at Bethesda Hospital, Yogyakarta, Indonesia.

There were 180 acute ischemic stroke patients who fulfilled the inclusion and exclusion criteria. Each subject recruited from acute stroke intensive care unit had been followed up from the first day they were hospitalized until hospital discharge (died or discharged alive) and 30 days after the onset.

Ethical approval number 1087/C.16/FK/2019 was obtained from Health Research Ethics Committee, Faculty of Medicine Duta Wacana Christian University Yogyakarta. This research has been registered at Center for Health Resources and Services Research and Development Indonesia with the ethical approval number of 1087/C.16/FK/2019.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Adult age (>18 years old)
* Diagnosed with acute ischemic stroke for the first time
* The onset is <24 hours
* Not a referral patient
* GCS score of 15 (fully alert)
* Mild to moderate scores on NIHSS

Exclusion Criteria:

* Subjects known to have hypersensitivity to DLBS1033
* Participated in other studies for the past 1 month
* Not competent enough in giving approval and answering questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Improvement in modified Rankin Scale (mRS) scores at hospital discharge | At hospital discharge (approximately 4 days after treatment initiation)
  Change in functional outcomes as measured by Modified Rankin Scale (MRS) from its baseline value.
Improvement in modified Rankin Scale (mRS) scores at 30 days | 30 days after treatment initiation
  Change in functional outcomes as measured by Modified Rankin Scale (MRS) from its hospital discharge value.
Improvement in National Institutes of Health Stroke Scale (NIHSS) scores at hospital discharge | At hospital discharge (approximately 4 days after treatment initiation)
  Change in functional outcomes as measured by National Institutes of Health Stroke Scale (NIHSS) from its baseline value.
Improvement in National Institutes of Health Stroke Scale (NIHSS) scores at 30 days | 30 days after treatment initiation
  Change in functional outcomes as measured by National Institutes of Health Stroke Scale (NIHSS) from its hospital discharge value.
Improvement in Barthel Index (BI) scores at hospital discharge | At hospital discharge (approximately 4 days after treatment initiation)
  Change in functional outcomes as measured by Barthel Index (BI) from its baseline value.
Improvement in Barthel Index (BI) scores at 30 days | 30 days after treatment initiation
  Change in functional outcomes as measured by Barthel Index (BI) from its hospital discharge value.

CONTACTS AND LOCATIONS:
Overall Officials: Rizaldy Pinzon, MD, MSc, PhD, Principal Investigator — Duta Wacana Christian University
Locations (1):
- Bethesda Hospital Yogyakarta, Yogyakarta, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krishnamurthi RV, Feigin VL, Forouzanfar MH, Mensah GA, Connor M, Bennett DA, Moran AE, Sacco RL, Anderson LM, Truelsen T, O'Donnell M, Venketasubramanian N, Barker-Collo S, Lawes CM, Wang W, Shinohara Y, Witt E, Ezzati M, Naghavi M, Murray C; Global Burden of Diseases, Injuries, Risk Factors Study 2010 (GBD 2010); GBD Stroke Experts Group. Global and regional burden of first-ever ischaemic and haemorrhagic stroke during 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet Glob Health. 2013 Nov;1(5):e259-81. doi: 10.1016/S2214-109X(13)70089-5. Epub 2013 Oct 24. PMID 25104492
- [Background] Mellor RM, Bailey S, Sheppard J, Carr P, Quinn T, Boyal A, Sandler D, Sims DG, Mant J, Greenfield S, McManus RJ. Decisions and delays within stroke patients' route to the hospital: a qualitative study. Ann Emerg Med. 2015 Mar;65(3):279-287.e3. doi: 10.1016/j.annemergmed.2014.10.018. Epub 2014 Nov 15. PMID 25455907
- [Background] Ogbole GI, Owolabi MO, Ogun O, Ogunseyinde OA, Ogunniyi A. TIME OF PRESENTATION OF STROKE PATIENTS FOR CT IMAGING IN A NIGERIAN TERTIARY HOSPITAL. Ann Ib Postgrad Med. 2015 Jun;13(1):23-8. PMID 26807083
- [Background] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265
- [Background] Tjandrawinata RR, Trisina J, Rahayu P, Prasetya LA, Hanafiah A, Rachmawati H. Bioactive protein fraction DLBS1033 containing lumbrokinase isolated from Lumbricus rubellus: ex vivo, in vivo, and pharmaceutic studies. Drug Des Devel Ther. 2014 Sep 25;8:1585-93. doi: 10.2147/DDDT.S66007. eCollection 2014. PMID 25284988
- [Background] Toyoda K. Epidemiology and registry studies of stroke in Japan. J Stroke. 2013 Jan;15(1):21-6. doi: 10.5853/jos.2013.15.1.21. Epub 2013 Jan 31. PMID 24324936
- [Background] Trisina J, Sunardi F, Suhartono MT, Tjandrawinata RR. DLBS1033, a protein extract from Lumbricus rubellus, possesses antithrombotic and thrombolytic activities. J Biomed Biotechnol. 2011;2011:519652. doi: 10.1155/2011/519652. Epub 2011 Mar 3. PMID 21403877
- [Background] Venketasubramanian N, Yoon BW, Pandian J, Navarro JC. Stroke Epidemiology in South, East, and South-East Asia: A Review. J Stroke. 2017 Sep;19(3):286-294. doi: 10.5853/jos.2017.00234. Epub 2017 Sep 29. PMID 29037005
- [Background] Zhou M, Offer A, Yang G, Smith M, Hui G, Whitlock G, Collins R, Huang Z, Peto R, Chen Z. Body mass index, blood pressure, and mortality from stroke: a nationally representative prospective study of 212,000 Chinese men. Stroke. 2008 Mar;39(3):753-9. doi: 10.1161/STROKEAHA.107.495374. Epub 2008 Jan 31. PMID 18239175